CLINICAL TRIAL: NCT01064791
Title: A Partially Blinded, Prospective, Randomized Multicenter Study Evaluating Efficacy, Safety and Tolerability of Oral Sotrastaurin Plus Standard or Reduced Exposure Tacrolimus vs. Mycophenolic Acid Plus Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Sotrastaurin Combined With Tacrolimus vs. a Mycophenolic Acid-tacrolimus Regimen in Renal Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAEB071A2214; 2009-015456-14 (EudraCT Number)
Record Dates: First submitted 2010-02-02; First posted 2010-02-08 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2016-11

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation
MeSH Terms: interventions — sotrastaurin; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm 1 (Experimental): sotrastaurin (100mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (Dose 1) + tacrolimus + standard of care medications
- Arm 2 (Experimental): sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (Dose 2) + tacrolimus + standard of care medications
- Arm 3 (Experimental): sotrastaurin (300mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: sotrastaurin (Dose 3) + tacrolimus + standard of care medications
- Arm 4 (Active Comparator): mycophenolic acid (720mg bid) + tacrolimus + standard of care medications
  Interventions: Drug: mycophenolic acid + tacrolimus + standard of care medications

INTERVENTIONS:
Drug: sotrastaurin (Dose 1) + tacrolimus + standard of care medications — sotrastaurin (100mg bid) + tacrolimus + standard of care medications
  Arms: Arm 1
Drug: sotrastaurin (Dose 2) + tacrolimus + standard of care medications — sotrastaurin (200mg bid) + tacrolimus + standard of care medications
  Arms: Arm 2
Drug: sotrastaurin (Dose 3) + tacrolimus + standard of care medications — sotrastaurin (300mg bid) + tacrolimus + standard of care medications
  Arms: Arm 3
Drug: mycophenolic acid + tacrolimus + standard of care medications — mycophenolic acid (720mg bid) + tacrolimus + standard of care medications
  Arms: Arm 4

SUMMARY:
This study will assess the safety and efficacy of different doses of sotrastaurin when combined with tacrolimus for the prevention of acute rejection after de novo renal transplantation.

ELIGIBILITY:
Inclusion criteria:

* Recipients of a first or second kidney transplant from a deceased, living unrelated or non-human leukocyte antigen (HLA) identical living related donor.
* Recipients of a kidney with a cold ischemia time < 30 hours.
* Recipients of a kidney from a donor 10 - 65 years old.

Exclusion criteria:

* Multi-organ transplant recipients.
* Recipients of an organ from an non-heart beating donor.
* Patients receiving a second kidney allograft if the first allograft was
* Functional for less than three years
* Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) at screening and cannot discontinue this treatment.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Demonstrate that at least one of the sotrastaurin + tacrolimus treatment arms is non-inferior to the active control regimen with respect to composite efficacy failure (treated BPAR of grade IA or higher, graft loss, death or lost to follow up). | Month 6

SECONDARY OUTCOMES:
Evaluate renal allograft function post-transplantation (estimated GFR by MDRD equation; estimated creatinine clearance by Cockroft-Gault formula; serum creatinine) | Months 6, 12, 24, and 36
Demonstrate that at least one of the sotrastaurin + tacrolimus treatment arms is non-inferior to the active control regimen with respect to composite efficacy failure (treated BPAR of grade IA or higher, graft loss, death or lost to follow up). | Months 12, 24, and 36
Evaluate individual components of the composite efficacy endpoint (treated BPAR, severity of acute rejections by Banff 2007 diagnostic category). | Months 6, 12, 24, and 36
Evaluate safety and tolerability (adverse events, serious adverse events, laboratory abnormalities, vital signs, electrocardiograms, physical examination). | Months 6, 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmceuticals, Study Director — Novartis Pharmceuticals
Locations (39):
- United States (6):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Madison, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
- Australia (4):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- Novartis Investigative Site, Cali, Colombia
- Novartis Investigative Site, Aarhus, Denmark
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Regensburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Rotterdam, Netherlands
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Seoul, Korea, South Korea
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Manchester

REFERENCES:
- [Result] Russ GR, Tedesco-Silva H, Kuypers DR, Cohney S, Langer RM, Witzke O, Eris J, Sommerer C, von Zur-Muhlen B, Woodle ES, Gill J, Ng J, Klupp J, Chodoff L, Budde K. Efficacy of sotrastaurin plus tacrolimus after de novo kidney transplantation: randomized, phase II trial results. Am J Transplant. 2013 Jul;13(7):1746-56. doi: 10.1111/ajt.12251. Epub 2013 May 13. PMID 23668931
- See also: Novartis Results on CAEB071A2214 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10063